CLINICAL TRIAL: NCT01458821
Title: Investigating the Impact of Cognitive Training for Firefighters With Tinnitus
Brief Title: Cognitive Training for Firefighters With Tinnitus
Acronym: FEMAICT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Federal Emergency Management Agency (U.S. Federal Agency)
Responsible Party: Principal Investigator, Jay F. Piccirillo, MD, Professor, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201110046; EMW-2010-FP-00601 (Other Grant/Funding Number: FEMA Assistance to Firefighters Grant Program)
Record Dates: First submitted 2011-10-10; First posted 2011-10-25 (Estimated); Last update posted 2014-05-09 (Estimated); Status verified 2014-05

CONDITIONS: Tinnitus
Keywords: Tinnitus
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Brain Fitness Program - Tinnitus (Experimental): Brain Fitness Program-Tinnitus was developed to improve cognitive function by engaging the brain's neuroplasticity; the program is novel, non-invasive, and inexpensive.
  Interventions: Behavioral: Brain Fitness Program - Tinnitus
- No treatment (No Intervention): Subject will make no changes in their usual daily routine. No intervention. Will repeat all study procedures at end of 8 weeks.

INTERVENTIONS:
Behavioral: Brain Fitness Program - Tinnitus — Brain Fitness Program-Tinnitus was developed to improve cognitive function by engaging the brain's neuroplasticity; the program is novel, non-invasive, and inexpensive.
  Other Names: Posit Science
  Arms: Brain Fitness Program - Tinnitus

SUMMARY:
The purpose of this research study is to determine whether the Brain Fitness Program-Tinnitus affects how tinnitus is perceived and if its use aids in the recovery of cognitive functions that may be affected by tinnitus. The investigators hope to better understand areas of the brain involved with or changed because of tinnitus. The investigators also hope to see if the Brain Fitness Program-Tinnitus impacts changes in those areas of the brain the investigators believe may be affected by tinnitus.

DETAILED DESCRIPTION:
The objective of this pilot research project is to advance knowledge about the role of attention, control, and other cortical networks in the development and maintenance of bothersome tinnitus.

The investigators have three specific aims. First, determine whether the Brain Fitness Program-Tinnitus affects the tinnitus percept and aids the recovery of cognitive functions apparently "highjacked" by the tinnitus. Brain Fitness Program-Tinnitus was developed to improve cognitive function by engaging the brain's neuroplasticity; the program is novel, non-invasive, and inexpensive. Second, establish specific default mode, attention system, and cognitive control network deficits in patients with bothersome tinnitus through the use of advanced neuroimaging techniques. Third, assess whether exposure to the Brain Fitness Program-Tinnitus impacts changes in the default mode, attention system, and cognitive control network deficits.

The investigators will employ a randomized clinical trial design among a cohort of active-duty firefighters who experience bothersome tinnitus. A planned enrollment of 40 firefighters with tinnitus in the clinical trial will have sufficient statistical power to detect a 17-point change in Tinnitus Handicap Inventory scores. In addition, a previously developed fcMRI protocol will be used to study brain activity in regions associated with voluntary, involuntary, and executive control of attention in 60 firefighters (40 firefighters enrolled in the clinical trial and 20 firefighters without tinnitus).

ELIGIBILITY:
Inclusion Criteria:

* Able to give informed consent
* Men and women between the ages of 20 and 65 years
* Must be able to read, write, and understand English
* Subjective, unilateral or bilateral, non-pulsatile tinnitus of 6 month's duration or greater
* Score of 3, 4, or 5 on the Global Bothersome scale
* Have access to uninterrupted use of computer in quiet setting for minimum of 1 hour per day/5 days per week for 2 months.
* Be willing to be randomized to either arm of the study.

Exclusion Criteria:

* Currently taking medication for depression, anxiety, or other DSM IV Axis 1 disorder
* History of head trauma sufficient to cause loss of consciousness for ≥30 minutes
* History of surgery to the brain
* History of claustrophobia, which will prevent subject from completing MRI
* Presence of metallic implants in the head and upper cervical region that are non-MRI compatible and would prohibit use of MRI
* Patients with cardiac pacemakers, intracardiac lines, implanted medication pumps, implanted electrodes in the brain, or any other contraindication for MRI scan
* Currently pregnant
* Patients with an acute or chronic unstable medical condition, which, in the opinion of the investigator, would prevent them from successfully participating in the study
* Patients with any active ear disease, which, in the opinion of the PI, needs to be further evaluated
* Patients with symptoms of depression as evidenced by a score of 15 or greater on the PHQ-9
* Any psychiatric co-morbidity that may complicate the interpretation of study results
* History of seizure disorder or any other neurological condition
* Weight over 350 pounds
* Inability to lay flat for 2 hours
* Active alcohol and/or drug dependence or history of alcohol and/or drug dependence within the last year
* Any medical condition, which, in the opinion of the PI, confounds study results or places the subject at greater risk
* Prior use of Posit Science Brain Fitness Program, or any other cognitive training program (regular or tinnitus) in the past year
* Patients with hyperacusis (hyper-sensitivity to noises) or misophonia (abnormally strong reactions of the autonomic and limbic systems to sound)
* Tinnitus related to cochlear implantation, retrocochlear lesion, Meniere's Disease, or other known anatomic lesions of the ear or temporal bone
* Tinnitus related to a Workman's Compensation claim or litigation-related event that is still pending.
* History of irritable bowel syndrome, fibromyalgia, chronic fatigue syndrome, or other illnesses or disorders that falls into the category of functional somatic syndromes.(Barsky and Borus 1999)

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-03; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Tinnitus Handicap Inventory at 8 weeks post Brain Fitness use. | 8 weeks.
  Patient-based rating scale of tinnitus severity

SECONDARY OUTCOMES:
Change in Baseline Tinnitus Bother Score at 8 weeks post Brain Fitness Program Use. | 8 weeks
  Neuropsychological test to assess an individual's verbal learning and memory abilities

CONTACTS AND LOCATIONS:
Overall Officials: Jay F Piccirillo, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Derived] Kallogjeri D, Piccirillo JF, Spitznagel E Jr, Hale S, Nicklaus JE, Hardin FM, Shimony JS, Coalson RS, Schlaggar BL. Cognitive Training for Adults With Bothersome Tinnitus: A Randomized Clinical Trial. JAMA Otolaryngol Head Neck Surg. 2017 May 1;143(5):443-451. doi: 10.1001/jamaoto.2016.3779. PMID 28114646